CLINICAL TRIAL: NCT00598832
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study to Demonstrate the Efficacy and Safety of Adapalene Lotion, 0.1% Compared With Vehicle Lotion in Subjects With Acne Vulgaris
Brief Title: Clinical Study to Test the Efficacy and Safety of Adapalene, 0.1%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Marie Ciardella Clinical Trials.gov Administrator, Galderma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18113; IND 076057
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-03

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Adapalene
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapalene lotion 0.1% (Experimental)
  Interventions: Drug: Adapalene lotion 0.1%
- Adapalene Lotion vehicle (Placebo Comparator)
  Interventions: Drug: Adapalene Lotion Vehicle

INTERVENTIONS:
Drug: Adapalene lotion 0.1% — Adapalene, 0.1% will be applied topically to the face, once a day, for 12 weeks
  Arms: Adapalene lotion 0.1%
Drug: Adapalene Lotion Vehicle — Adapalene Lotion Vehicle will be applied topically to the face, once a day, for 12 weeks
  Arms: Adapalene Lotion vehicle

SUMMARY:
The purpose of this study is to determine whether Adapalene, 0.1% is safe and effective in the treatment of Acne Vulgaris.

DETAILED DESCRIPTION:
This study will compare the efficacy and safety of Adapalene, 0.1% and vehicle in the treatment of subjects with Acne Vulgaris. This is a multi-center, randomized, double-blind, parallel, vehicle controlled study involving subjects with acne vulgaris meeting pre-specified inclusion/exclusion criteria. Male and female subjects, 12 years of age or older, with 20-50 papules and pustules and 30 to 100 non-inflammatory lesions and have an Investigator's Global Assessment (IGA) score of 3 (Moderate) or 4 (Severe) are eligible for enrollment. One nodule may be present at inclusion. Acne lesions are evaluated on the face only. Subjects presenting with facial and truncal acne vulgaris can participate in this study. Subjects will be randomized in a 1:1 ratio to Adapalene, 0.1% or Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Moderate or Severe Acne Vulgaris,
* 20-50 papules and pustules in total on the face excluding the nose
* 30-100 non-inflammatory lesions on the face excluding the nose.
* Negative urine pregnancy test for all females.

Exclusion Criteria:

* Subjects with more than one acne nodule.
* Subjects with any acne cyst on the face.
* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), or severe acne requiring systemic treatment.
* Subjects with underlying diseases or other dermatologic conditions that require the use of interfering topical or systemic therapy, such as, but not limited to, atopic dermatitis, perioral dermatitis or rosacea.
* Subjects who are pregnant, nursing, or planning a pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (27):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Scott Dinehart, Little Rock, Arkansas
  - Dermatology and Laser Center, Marina del Rey, California
  - Therapeutics Clinical Research, San Diego, California
  - Solano Clinical Research, Vallejo, California
  - Colorado Medical Research Center, Denver, Colorado
  - Longmont Clinic, Longmont, Colorado
  - Advanced Dermatology, Clermont, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Anne M. Loebl, Augusta, Georgia
  - Scott Glazer, Buffalo Grove, Illinois
  - Sound Bend Clinic, South Bend, Indiana
  - Hamzavi Dermatology, Port Huron, Michigan
  - Central Dermatology, PC, St Louis, Missouri
  - Darmouth-Hitchcock Medical Center Section of Dermatology, Lebanon, New Hampshire
  - Academic Dermatology, Albuquerque, New Mexico
  - Elizabeth Arthur, Rochester, New York
  - Derm Research Center of New York, Stony Brook, New York
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Haber Dermatology & Cosmetic Research, South Euclid, Ohio
  - OU Health Sciences Center-Dept. of Dermatology, Oklahoma City, Oklahoma
  - Oregon Medical Center, PC, Portland, Oregon
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Center for Clinical Studies, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (7):
  - The Dermatology Centre, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Dermadvance Research, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Lynderm Research, Inc., Markham, Ontario
  - K. Papp Clinical Research, Inc., Waterloo, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi center study recruitment period: First subject enrolled Nov 7, 2007; last subject completed Nov 6, 2008
Pre-assignment Details: Washout requirements: 2 weeks for systemic anti-inflammatory drugs, 4 weeks for oral antibiotics, 2 months for inhaled/nasal steroids and 6 months for hormonal contraceptives/therapies.
Groups:
- Adapalene Lotion 0.1%; Adapalene Lotion Vehicle 0%: once a day for 12 weeks
Period: Overall Study
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Started | 533 | 542
Completed | 471 | 460
Not Completed | 62 | 82
Not completed — Lack of Efficacy | 3 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 25 | 36
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 24 | 29
Not completed — Pregnancy | 2 | 2
Not completed — Physician Decision | 1 | 4
Not completed — Non compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0% | Total
Number analyzed (Participants) | 533 | 542 | 1075
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 327 | 343 | 670
  Between 18 and 65 years | 206 | 199 | 405
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (7.1) | 18.9 (6.5) | 19.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283 | 290 | 573
  Male | 250 | 252 | 502
Region of Enrollment [Number; unit: participants]
  United States | 463 | 468 | 931
  Canada | 70 | 74 | 144

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Endpoint: Success Rate on Investigator's Global Assessment (IGA) From Baseline to Week 12
Description: Success defined as percentage of subjects who achieved at least a two-grade reduction in IGA scale (e.g from moderate to clear or almost clear)at week 12 from baseline, Last Observation Carried Forward, Intent to treat population. The IGA (Investigator Global Assessment) is defined as a 5 point scale (0 to 4). "0" = clear , "1"= almost clear, "2"= mild, "3"= moderate, "4"=severe.
Time Frame: From Baseline to Week 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 533 | 542
Percentage of Participants | 26.3 | 17.3

2. Secondary Outcome: Mean Percent Change in Total Lesion Count From Baseline to Week 12
Description: Percent change in lesion count from baseline to week 12
Time Frame: From Baseline to Week 12
Measure: Mean (Standard Deviation); unit: % Change in Lesion Count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 533 | 542
% Change in Lesion Count
  Total lesion count | -51.5 (29.6) | -37.1 (34.2)
  Inflammatory | -54.9 (31.9) | -40.3 (40.7)
  Non-Inflammatory | -49.6 (34.0) | -35.7 (38.0)

3. Primary Outcome: Co-Primary Endpoint: Absolute Change in Total Lesion Count From Baseline to Week 12
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Total Lesion Count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 533 | 542
Absolute Change in Total Lesion Count | 36.7 (1.0) | 25.5 (1.0)

4. Primary Outcome: Co-Primary Endpoint: Absolute Change in Inflammatory Lesion Count From Baseline to Week 12
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Infl Lesion count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 533 | 542
Absolute Change in Infl Lesion count | 14.3 (0.4) | 10.2 (0.4)

5. Primary Outcome: Co-Primary Endpoint: Absolute Change in NonInflammatory Lesion Counts From Baseline to Week 12
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: Absolute Change in Non-Infl Lesion count
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Number analyzed (Participants) | 533 | 542
Absolute Change in Non-Infl Lesion count | 22.4 (0.8) | 15.3 (0.7)

ADVERSE EVENTS:
Arm/Group | Adapalene Lotion 0.1% | Adapalene Lotion Vehicle 0%
Serious Adverse Events (participants affected / at risk) | 2/533 | 2/542
Other Adverse Events (participants affected / at risk) | 50/533 | 21/542
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene Lotion 0.1% (N=533) | Adapalene Lotion Vehicle 0% (N=542)
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene Lotion 0.1% (N=533) | Adapalene Lotion Vehicle 0% (N=542)
Dry skin (Skin and subcutaneous tissue disorders) | 50 (50) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
disclosure restriction varies per institutional request/agreement